CLINICAL TRIAL: NCT05795153
Title: A Multicenter, Open-label Phase 3 Study: Ambulatory Blood Pressure Monitoring in Adult Patients With Chronic Spontaneous Urticaria Inadequately Controlled by H1-antihistamines Treated With Remibrutinib up to 12 Weeks.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLOU064A2305; 2022-002838-13 (EudraCT Number)
Record Dates: First submitted 2023-03-21; First posted 2023-04-03 (Actual); Results first posted 2025-04-30 (Actual); Last update posted 2025-10-16 (Actual); Status verified 2025-10

CONDITIONS: Chronic Spontaneous Urticaria
Keywords: Chronic Spontaneous Urticaria (CSU); remibrutinib; Systolic Blood Pressure (SBP); Diastolic Blood Pressure (DBP); Ambulator Blood Pressure Monitoring (ABPM); H1 antihistamines (H1-AH) treatment
MeSH Terms: conditions — Chronic Urticaria | interventions — remibrutinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- LOU064 (remibrutinib) (Experimental): All participants were assigned to remibrutinib 25 mg b.i.d. for 12 weeks.
  Interventions: Drug: LOU064

INTERVENTIONS:
Drug: LOU064 — One film-coated tablet (25 mg) was to be taken in the morning and evening, respectively, with a 12-hour interval at approximately the same time everyday.
  Other Names: remibrutinib

SUMMARY:
The purpose of this study was to assess the effect of remibrutinib 25 mg twice a day (b.i.d.) open-label on Systolic Blood Pressure (SBP) measured as a change in 24-hour weighted average SBP from baseline to Week 4 assessed by Ambulator Blood Pressure Monitoring (ABPM); and to assess overall safety and efficacy over 12 weeks in adult participants with Chronic Spontaneous Urticaria (CSU) inadequately controlled with second generation H1 antihistamines (H1-AH) treatment. ABPM was chosen for the blood pressure assessment in this trial as recommended by the FDA for drugs intended for chronic use (Assessment of Pressor Effects of Drugs Guidance for Industry (FDA 2022)).

DETAILED DESCRIPTION:
This study consisted of a screening period of up to 4 weeks, a 12-week open-label treatment period and a treatment-free follow-up period of 4 weeks, with a total study duration of up to 20 weeks.

At the end of the treatment phase, participants had the option to continue in an extension study (CLOU064A2303B (NCT05513001)) if approved in the country and at the site.

ELIGIBILITY:
Key Inclusion Criteria:

* Signed informed consent obtained prior to participation in the study
* Male and female adult participants >= 18 years of age
* CSU duration for >= 6 months prior to screening (defined as the onset of CSU determined by the Investigator based on all available supporting documentation).
* Diagnosis of CSU inadequately controlled by second generation H1-AH at the time of baseline (Day 1)
* Documentation of hives within three months before baseline (either at screening and/or at baseline (Day 1); or documented in the participants' medical history).
* Willing and able to complete an Urticaria Patient Daily Diary (UPDD) for the duration of the study and adhere to the protocol
* Participants had no more than 2 missing UPDD entries (either morning or evening) in the 7 days prior to baseline (Day 1).

Key Exclusion Criteria:

* Participants unable to tolerate 24-hour ambulatory blood pressure measurement using automatic ABPM device
* Ongoing or past history of hypertension and/or SBP >= 140 or =< 90 OR DBP >= 90 or =< 60 mmHg at screening
* Participants working night shifts
* Participants taking/requiring medications prohibited by the protocol (including those known to interfere with blood pressure assessments in the study)
* Evidence of clinically significant cardiovascular, neurological, psychiatric, pulmonary, renal, hepatic, endocrine, metabolic, hematological disorders, gastrointestinal disease or immunodeficiency that, in the Investigator's opinion, would compromise the safety of the participant, interfere with the interpretation of the study results or otherwise preclude participation or protocol adherence of the participant.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Actual)
Dates: Start 2023-04-05 (Actual); Primary Completion 2024-04-25 (Actual); Study Completion 2024-04-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (43):
- United States (10):
  - Acuro Research Inc, Little Rock, Arkansas
  - Florida Ctr Allergy Asthma Research, Aventura, Florida
  - Finlay Medical Research, Greenacres City, Florida
  - Treasure Valley Medical Research, Boise, Idaho
  - Endeavor Health, Glenview, Illinois
  - Allergy and Asthma Specialist P S C, Owensboro, Kentucky
  - Allergy Asthma and Clinical Research, Oklahoma City, Oklahoma
  - Allergy and Clinical Immunology Associates, Pittsburgh, Pennsylvania
  - Western Sky Medical Research, El Paso, Texas
  - Allergy Asthma and amp Sinus Ctr S C, Greenfield, Wisconsin
- Argentina (4):
  - Novartis Investigative Site, Nueve de Julio, Buenos Aires
  - Novartis Investigative Site, Sourigues, Buenos Aires
  - Novartis Investigative Site, Santa Fe, Rosario
  - Novartis Investigative Site, Rosario, Santa Fe Province
- Canada (2):
  - Novartis Investigative Site, Calgary, Alberta
  - Novartis Investigative Site, Montreal, Quebec
- France (8):
  - Novartis Investigative Site, Angers
  - Novartis Investigative Site, Antony
  - Novartis Investigative Site, Brest
  - Novartis Investigative Site, Montpellier
  - Novartis Investigative Site, Paris
  - Novartis Investigative Site, Reims
  - Novartis Investigative Site, Saint-Mandé
  - Novartis Investigative Site, Toulouse
- Germany (6):
  - Novartis Investigative Site, Bramsche, Lower Saxony
  - Novartis Investigative Site, Göttingen, Lower Saxony
  - Novartis Investigative Site, Halle, Saxony-Anhalt
  - Novartis Investigative Site, Erlangen
  - Novartis Investigative Site, Hanover
  - Novartis Investigative Site, Marburg
- Novartis Investigative Site, Singapore, Singapore
- Slovakia (3):
  - Novartis Investigative Site, Komárno
  - Novartis Investigative Site, Levice
  - Novartis Investigative Site, Nové Zámky
- South Korea (3):
  - Novartis Investigative Site, Daegu, Dalseo Gu
  - Novartis Investigative Site, Suwon, Gyeonggi-do
  - Novartis Investigative Site, Seoul
- Spain (3):
  - Novartis Investigative Site, Alicante, Valencia
  - Novartis Investigative Site, Valencia, Valencia
  - Novartis Investigative Site, Madrid
- Turkey (Türkiye) (3):
  - Novartis Investigative Site, Izmir
  - Novartis Investigative Site, Kayseri
  - Novartis Investigative Site, Samsun

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing access to patient-level data and supporting clinical documents from eligible studies with qualified external researchers. Requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to protect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

REFERENCES:
- See also: A Plain Language Trial Summary is available on www.novctrd.com — https://www.novctrd.com/ctrdweb/patientsummary/patientsummaries?patientSummaryId=2573

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted globally across 10 countries: Argentina (4 centers), Canada (2 centers), France (8 centers), Germany (6 centers), Republic of Korea (3 centers), Singapore (1 center), Slovakia (3 centers), Spain (4 centers), Turkey (3 centers), and USA (11 centers).
Pre-assignment Details: Participants underwent a screening period of up to 4 weeks.
Period: Overall Study
Arm/Group | LOU064 (Remibrutinib)
Started | 144
Completed | 137
Not Completed | 7
Not completed — Adverse Event | 2
Not completed — Unsatisfactory therapeutic effect | 2
Not completed — Lost to Follow-up | 1
Not completed — Subject decision | 2

BASELINE CHARACTERISTICS:
Arm/Group | LOU064 (Remibrutinib)
Number analyzed (Participants) | 144
Age, Continuous [Mean (Standard Deviation); unit: Years] | 42.2 (14.52)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 105
  Male | 39
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 19
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 89
  More than one race | 0
  Unknown or Not Reported | 32
Baseline Systolic Blood Pressure (SBP) [Mean (Standard Deviation); unit: millimeter of mercury (mmHg)] | 117.1 (13.11)
Baseline Diastolic Blood Pressure (DBP) [Mean (Standard Deviation); unit: millimeter of mercury (mmHg)] | 75.0 (8.98)

OUTCOME MEASURES:

1. Primary Outcome: Estimated Mean Change From Baseline at Week 4 in 24-hour Systolic Blood Pressure (SBP) Measured by Ambulatory Blood Pressure Monitoring (ABPM)
Description: A linear regression with SBP as a covariate was employed. The change in SBP from baseline to Week 4 was predicted at the median baseline level. The change from baseline in the 24-hour weighted average SBP was calculated using the time weighted average of the area under the curve (AUC) of SBP obtained over a 24-hour period as measured by ABPM. That is, the time weighted average of AUC of 24-hour SBP obtained at baseline was subtracted from corresponding time weighted average of AUC of SBP at Week 4.
  In the analysis, if participants took prohibited antihypertensive treatment before Week 4, their subsequent measurements were excluded. In such cases, the excluded measurements were imputed by increasing the 24-hour SBP by 3 mmHg from the baseline value at Week 4. Moreover, participants who discontinued of study treatment due to any reason prior to the Week 4 were excluded from the analysis. The Mixed Models for Repeated Measures (MMRM) approach was used.
Time Frame: Baseline, Week 4
Population: Full Analysis Set (FAS): all participants to whom study treatment was assigned and received at least one dose of treatment. Participants who discontinued treatment prior to Week 4 were excluded from the analysis.
Measure: Mean (95% Confidence Interval); unit: millimeter of mercury (mmHg)
Arm/Group | LOU064 (Remibrutinib)
Number analyzed (Participants) | 143
millimeter of mercury (mmHg) | -1.3 [-2.3 to -0.3]

2. Secondary Outcome: Observed Mean Change From Baseline to Week 4 in 24-hour Weighted Average Systolic Blood Pressure (SBP) Measured by ABPM
Description: The change from baseline in the 24-hour weighted average systolic blood pressure (SBP) was calculated using the time weighted average of the area under the curve (AUC) of SBP obtained over a 24-hour period as measured by ABPM. This analysis was conducted using the observed data.
  Data was computed taking weighted averages over time and discarding time intervals of more than 1 hour without measurements.
Time Frame: Baseline, Week 4
Population: Full Analysis Set (FAS): all participants to whom study treatment was assigned and received at least one dose of treatment. Only participants with a value at both baseline and Week 4 were included.
Measure: Mean (Standard Deviation); unit: millimeter of mercury (mmHg)
Arm/Group | LOU064 (Remibrutinib)
Number analyzed (Participants) | 142
millimeter of mercury (mmHg) | -1.65 (6.905)

3. Secondary Outcome: Estimated Mean Change From Baseline at Week 4 in 24-hour Diastolic Blood Pressure (DBP) Measured by ABPM
Description: A linear regression with DBP as a covariate was employed. The change in DBP from baseline to Week 4 was predicted at the median baseline level. The change from baseline in the 24-hour weighted average DBP was calculated using the time weighted average of the area under the curve (AUC) of DBP obtained over a 24-hour period as measured by ABPM. That is, the time weighted average of AUC of 24-hour DBP obtained at baseline was subtracted from corresponding time weighted average of AUC of DBP at Week 4.
  In the analysis, if participants took prohibited antihypertensive treatment before Week 4, their subsequent measurements were excluded. In such cases, the excluded measurements were imputed by increasing the 24-hour DBP by 3 mmHg from the baseline value at Week 4. Moreover, participants who discontinued of study treatment due to any reason prior to the Week 4 were excluded from the analysis. The Mixed Models for Repeated Measures (MMRM) approach was used.
Time Frame: Baseline, Week 4
Population: FAS: all participants to whom study treatment was assigned and received at least one dose of treatment. Participants who discontinued treatment prior to Week 4 were excluded from the analysis.
Measure: Mean (95% Confidence Interval); unit: millimeter of mercury (mmHg)
Arm/Group | LOU064 (Remibrutinib)
Number analyzed (Participants) | 143
millimeter of mercury (mmHg) | -0.1 [-0.8 to 0.6]

4. Secondary Outcome: Estimated Mean Change From Baseline at Week 4 in Daytime and Nighttime Average SBP Measured by ABPM
Description: The change in daytime (respectively nighttime) weighted average SBP was analyzed using linear regression model with baseline weighted average daytime SBP (respectively nighttime) as a covariate. The change in daytime (respectively nighttime) SBP from baseline to Week 4 was predicted at the median baseline level. The change from baseline of daytime (respectively nighttime) SBP was calculated using the time weighted average of the AUC of DBP obtained over daytime (respectively nighttime) In the analysis, if participants took prohibited antihypertensive treatment before Week 4, their subsequent measurements were excluded. In such cases, the excluded measurements were imputed by increasing the 24-hour SBP by 3 mmHg from the baseline value at Week 4. Moreover, participants who discontinued of study treatment due to any reason prior to the Week 4 were excluded from the analysis. The multiple imputation approach was used. Daytime: from 7am until 10 pm. Nighttime: from 10pm until 7 am.
Time Frame: Baseline, Week 4
Population: as for outcome 3
Measure: Mean (95% Confidence Interval); unit: millimeter of mercury (mmHg)
Arm/Group | LOU064 (Remibrutinib)
Number analyzed (Participants) | 143
millimeter of mercury (mmHg)
  daytime average SBP | -1.2 [-2.3 to -0.0]
  nighttime average SBP | -0.9 [-2.2 to 0.5]

5. Secondary Outcome: Estimated Mean Change From Baseline at Week 4 in Daytime and Nighttime Average DBP Measured by ABPM
Description: The change in daytime (respectively nighttime) weighted average DBP was analyzed using linear regression model with baseline weighted average daytime DBP (respectively nighttime) as a covariate. The change in daytime (respectively nighttime) DBP from baseline to Week 4 was predicted at the median baseline level. The change from baseline of daytime (respectively nighttime) DBP was calculated using the time weighted average of the AUC of DBP obtained over daytime (respectively nighttime) In the analysis, if participants took prohibited antihypertensive treatment before Week 4, their subsequent measurements were excluded. In such cases, the excluded measurements were imputed by increasing the 24-hour DBP by 3 mmHg from the baseline value at Week 4. Moreover, participants who discontinued of study treatment due to any reason prior to the Week 4 were excluded from the analysis. The multiple imputation approach was used. Daytime: from 7am until 10 pm. Nighttime: from 10pm until 7 am.
Time Frame: Baseline, Week 4
Population: as for outcome 3
Measure: Mean (95% Confidence Interval); unit: millimeter of mercury (mmHg)
Arm/Group | LOU064 (Remibrutinib)
Number analyzed (Participants) | 143
millimeter of mercury (mmHg)
  daytime average DBP | -0.6 [-1.3 to 0.2]
  nighttime average DBP | 0.2 [-0.8 to 1.1]

ADVERSE EVENTS:
Time Frame: On-treatment adverse events and deaths were reported from first dose of study medication up to 28 days after last dose of study medication, assessed up to approximately 18 weeks.
Description: Any sign or symptom that occurred during the conduct of the trial and safety follow-up. The safety analysis were done on the safety population, which included all enrolled subjects who received at least one dose of study medication.
Arm/Group | LOU064 (Remibrutinib)
All-Cause Mortality (participants affected / at risk) | 0/144
Serious Adverse Events (participants affected / at risk) | 4/144
Other Adverse Events (participants affected / at risk) | 32/144
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | LOU064 (Remibrutinib) (N=144)
Cholecystitis acute (Hepatobiliary disorders) | 1
Dizziness (Nervous system disorders) | 1
Chronic spontaneous urticaria (Skin and subcutaneous tissue disorders) | 1
Aortic dissection (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | LOU064 (Remibrutinib) (N=144)
Nasopharyngitis (Infections and infestations) | 12
Headache (Nervous system disorders) | 13
Chronic spontaneous urticaria (Skin and subcutaneous tissue disorders) | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2022-10-07): https://cdn.clinicaltrials.gov/large-docs/53/NCT05795153/Prot_000.pdf
  • Statistical Analysis Plan (2024-09-18): https://cdn.clinicaltrials.gov/large-docs/53/NCT05795153/SAP_001.pdf